CLINICAL TRIAL: NCT03478072
Title: The Role of Trichoscopy in the Preliminary Diagnosis of Immunobollous Diseases
Brief Title: Trichoscopy in Diagnosis of Immunobollous Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: tasbeeh salah (Other)
Responsible Party: Sponsor-Investigator, tasbeeh salah, principal investigator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: AUEC
Record Dates: First submitted 2018-03-15; First posted 2018-03-27 (Actual); Last update posted 2018-07-30 (Actual); Status verified 2018-07

CONDITIONS: IMMUNOBULLOUS DISEASES

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: trichoscopy — hair and scalp dermoscopy) is a non-invasive technique in which either a handheld dermoscope or a digital videodermoscope can be used to visualize hair and scalp structures

SUMMARY:
Autoimmune bullous diseases are a variety of skin diseases that are characterized by the presence of bullae or blisters. Most of these diseases are associated with substantial morbidity and mortality. They are classified according to the site of blister formation into intraepidermal as pemphigus valgaris and foliaceus, and subepidermal as bullous pemphigoid and dermatitis herpetiformis. These lesions commonly affect the scalp and manifest as blisters, erosions and crustations.

Trichoscopy (hair and scalp dermoscopy) is a non-invasive technique in which either a handheld dermoscope or a digital videodermoscope can be used to visualize hair and scalp structures. The method has well-established position as an ancillary tool in the diagnosis of many disorders such as, tinea capitis, alopecia areata, androgenetic alopecia, discoid lupus erythematosus, lichen planopilaris, folliculitis decalvans and other hair and scalp diseases. Few studies have reported that immunobullous diseases present characteristic trichoscopic patterns. So, Trichoscopy can be used as a rapid in-office preliminary diagnostic tool in the differential diagnosis of these diseases.

DETAILED DESCRIPTION:
Autoimmune bullous diseases are a variety of skin diseases that are characterized by the presence of bullae or blisters. Most of these diseases are associated with substantial morbidity and mortality. They are classified according to the site of blister formation into intraepidermal as pemphigus valgaris and foliaceus, and subepidermal as bullous pemphigoid and dermatitis herpetiformis. These lesions commonly affect the scalp and manifest as blisters, erosions and crustations.

Pemphigus is a group of potentially life-threatening intraepidermal vesiculobullous autoimmune diseases that affect the skin and mucous membranes. It is characterized by the presence of circulating and tissue-bound autoantibodies directed against desmogleins, which attaches adjacent epidermal cells via desmosomes. When autoantibodies attack desmogleins, the cells become separated from each other and the epidermis becomes "unglued", a phenomenon called acantholysis. This causes blisters that slough off and turn into sores.

In pemphigus vulgaris (PV) blisters and erosions occurs in the skin and/or mucous membranes, and circulating autoantibodies are directed against desmoglein 3 and 1. In pemphigus foliaceus, there is mainly skin involvement and antibodies are exclusively directed against desmoglein 1. Histologically, both subtypes exhibit intraepidermal blister formation with loss of keratinocytes' adhesion. However, in Pemphigus vulgaris, the split occurs just above the basal cell layer, whereas in pemphigus foliaceus it occurs in the upper part of the epidermis, at the level of the granular layer.

Bullous pemphigoid (BP) is a chronic, autoimmune, subepidermal, blistering skin disease that rarely involves mucous membranes. It is characterized by the presence of immunoglobulin G (IgG) autoantibodies specific for the hemidesmosomal BP antigens BP230 (BPAg1) and BP180 (BPAg2). The lesions of BP may initially start as an urticarial eruption, which over a course of weeks to months, develops into bullae. The lesions are usually prurutic. Once formed, blisters are large and tense, with a round or oval shape. Discrete lesions arise on normal or erythematous skin and are scattered throughout the body.

Dermatitis herpetiformis (DH) is an autoimmune blistering disorder associated in most patients with a gluten-sensitive enteropathy (GSE). DH is characterized by pruritic erythematous clusters of multiforme lesions, frequently in herpetiform pattern. Histopathologically, there are neutrophilic micro-abscesses in dermal papillae, dermal infiltration of neutrophils and eosinophils, and the formation of subepidermal vesicles. Blisters form within the lamina lucida.

Diagnosis of these diseases is based on clinical, histopathological, immunofluorescence and immunoserological tests. Because of the limited resources in our institution, diagnosis relies mainly on clinical and histopathological evaluations.

Trichoscopy (hair and scalp dermoscopy) is a non-invasive technique in which either a handheld dermoscope or a digital videodermoscope can be used to visualize hair and scalp structures. The method has well-established position as an ancillary tool in the diagnosis of many disorders such as, tinea capitis, alopecia areata, androgenetic alopecia, discoid lupus erythematosus, lichen planopilaris, folliculitis decalvans and other hair and scalp diseases. Few studies have reported that immunobullous diseases present characteristic trichoscopic patterns. So, Trichoscopy can be used as a rapid in-office preliminary diagnostic tool in the differential diagnosis of these diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical & histopathological diagnosis of autoimmune bullous diseases.

Exclusion Criteria:

* Patients who will not consent.
* Patients with any concomitant dermatological diseases.
* Pregnancy and lactation.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: upper Egyptian patients
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
trichoscopic features of autoimmune bullous diseases and frequency of each feature. | 1year
  Detect trichoscopic features of autoimmune bullous diseases and frequency of each feature.
diagnostic accuracy of trichoscopy in autoimmune bullous diseases. | 1year
  detect diagnostic accuracy of trichoscopy in autoimmune bullous diseases..

CONTACTS AND LOCATIONS:
Overall Officials: Nagwa Easa, prof, Study Chair — prof

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sar-Pomian M, Rudnicka L, Olszewska M. Trichoscopy - a useful tool in the preliminary differential diagnosis of autoimmune bullous diseases. Int J Dermatol. 2017 Oct;56(10):996-1002. doi: 10.1111/ijd.13725. Epub 2017 Aug 30. PMID 28856676
- [Result] Sar-Pomian M, Kurzeja M, Rudnicka L, Olszewska M. The value of trichoscopy in the differential diagnosis of scalp lesions in pemphigus vulgaris and pemphigus foliaceus. An Bras Dermatol. 2014 Nov-Dec;89(6):1007-12. doi: 10.1590/abd1806-4841.20143830. PMID 25387515